CLINICAL TRIAL: NCT04104217
Title: Music Therapy With Oncology Patients and Delirium: An Exploratory Study
Brief Title: A Study of the Experience of Music Therapy in Cancer Patients With Delirium
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: New York University (Other)
Responsible Party: Sponsor
Other Study IDs: 19-270
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Cancer Patients With Delirium
Keywords: Music therapy; 19-270
MeSH Terms: interventions — Music Therapy; Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- patients: Participate in 30-60 minute interviews after each music therapy session.
  Interventions: Behavioral: Music therapy; Behavioral: Interviews
- caregivers: Participate in 30-60 minute interviews after each music therapy session (ideally within 3 days).
  Interventions: Behavioral: Music therapy; Behavioral: Interviews
- nurses: Participate in 10-15 minute interviews after initial music therapy session.
  Interventions: Behavioral: Music therapy; Behavioral: Interviews
- music therapists: Music therapist will notify the researcher if he/she has provided music therapy for a patient who is identified as having delirium. Music therapists will also be interviewed about the clinical process after initial and follow up music sessions.
  Interventions: Behavioral: Interviews

INTERVENTIONS:
Behavioral: Music therapy — Music therapy sessions may last 20-60 minutes, with length and frequency to be determined mutually (generally 1-3 times per week). Music therapy sessions are done at the patient's bedside, where the music therapist plays live music on a guitar, keyboard, harp, or percussion instrument, sometimes as accompaniment to singing.
  Groups: caregivers; nurses; patients
Behavioral: Interviews — Each interview will be conducted in person in a private setting (with the exception of caregivers, who have the option to conduct interviews over the phone if it is not feasible to take place in the hospital). Each interview will follow a semi-structured interview guide and will ask for consent to audio record the interviews .

SUMMARY:
The purpose of this study is to improve our understanding of the experience of music therapy by cancer patients with delirium, and the experience of music therapists working with these patients. The researchers are focusing on patients with delirium because of the challenging symptoms of this condition.

At MSK, music therapy is routinely used in patients with cancer. Music therapy sessions are done at the patient's bedside, where the music therapist plays live music on a guitar, keyboard, harp, or percussion instrument, sometimes as accompaniment to singing.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (ages 18-75) with delirium
* referred for and receive music therapy.
* were identified as having delirium by the Confusion Assessment Method (CAM), Confusion Assessment Method for ICU patients (CAM-ICU) or a documented diagnosis by a clinician from the Department of Psychiatry and Behavioral Sciences in the patient's electronic medical record (EMR).
* Patients that have had music therapy in the past will be eligible for the study
* Only patients that recover from delirium (per CAM, CAM-ICU, or progress note by a clinician from the Department of Psychiatry and Behavioral Sciences) after receiving music therapy will be approached for interview by the researcher.

This study will also include their caregivers, music therapists, primary nurse, and bedside companions who have participated in or observed the participants' response to music therapy.

The music therapist participants are:

* Board-certified senior music therapists with 10 or more years experience in the research site who sign a blanket consent form to participate in study.
* Assigned to eligible patients by Integrative Medicine Service Client Service Representative (CSR).

The caregivers are:

* Family or unrelated adult (>18) caregivers who observed bedside music therapy session(s) with patients meeting inclusion criteria

The staff caregivers are:

* Primary nurse caring for eligible patients who receive their first music therapy session while experiencing delirium.
* Patient care technicians (PCT) assigned as bedside companions for eligible patients who receive music therapy

Exclusion Criteria:

* have a known hearing impairment
* do not speak English.
* are heavily sedated, comatose, or expected to be discharged or expire within 48 hours
* have known comorbidities of delirium tremens, steroid psychosis, or dementia

Caregivers will be excluded from the study if they do not speak English. Music therapists, nurses, or bedside companions will be excluded if they are not assigned to eligible patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient subjects who are referred for music therapy will be identified to the researcher by a board-certified music therapist on staff at MSKCC (excluding the Principal Investigator).
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
thematic analysis of data with music therapists | 1 year
  by interviews

SECONDARY OUTCOMES:
thematic analysis of data with caregivers, nurses, and patients | 1 year
  by interviews

CONTACTS AND LOCATIONS:
Overall Officials: Holly Mentzer, MA, LCAT, MT-BC, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm